CLINICAL TRIAL: NCT04552834
Title: Alterations of the Microbiome During Critical Illness With Short and Long Term Clinical Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1102
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Microbiome
Keywords: short term outcomes; long term outcomes
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to study the variations in the microbiome among critically ill patients and the effect of admission to the medical intensive care unit (MICU) at the University of Chicago. Additionally, investigators will examine the downstream clinical effects of dysbiosis in ICU patients and how patients maybe effected long term.

DETAILED DESCRIPTION:
During this study investigators will longitudinally collect discarded stool biosamples throughout the MICU admission when available. Stool Bio specimens will be recorded/coded and processed by the investigators. Stool Bio specimens will be analyzed for 16sRNA and metabolomics. Surveys will be conducted at study entry, in addition to 6 months and 12 months following discharge.

By longitudinally sampling discarded biospecimens from subjects throughout their MICU admission in additionally to describing long term following up. We will be able to correlate changes in the microbiome with clinical data, and follow up surveys to identify factors that may impact the composition of the microbiome and their impact on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

adult patients admitted to the intensive care unit

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients admitted to the intensive care unit
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Long Term Mortality | up to 1 year
  Death from any cause 90 day, 1 year

SECONDARY OUTCOMES:
hospital mortality | 28 day
  death from any cause during hospitalization
ICU length of stay | hospitalization up to 6 weeks
  number of days admitted to the ICU
Hospital length of stay | hospitalization up to 6 weeks
  number of days admitted to the hospital
Functional Status Score | up to 12 months after discharge
  Katz Index of Independence in activities of daily living; minimal score = 0; maximum score = 6; higher score better outcome
Cognitive Dysfunction | Up to 12 months after discharge
  Montreal Cognitive Assessment (MoCA) score; minimal score = 0; maximum score = 30; higher score better outcome
Quality of Life score | up to 12 months after discharge
  SF-36 score: including physical component summary (PCS) and mental component summary (MCS)

OTHER OUTCOMES:
ICU re-admission | up to 12 months
  number of admissions to ICU
ICU related complications | up to 6 weeks
  presence of ICU complications: including ventilator associated pneumonia, GI hemorrhage, DVT/PE, sacral decubitus ulcer, delirium, ICU acquired weakness
Ventilator days | up to 4 weeks
  duration of mechanical ventilation via endotracheal tube

CONTACTS AND LOCATIONS:
Overall Officials: Bhakti Patel, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States